CLINICAL TRIAL: NCT04100018
Title: A Phase 3, Randomized, Double-Blind Study of Nivolumab or Placebo in Combination With Docetaxel, in Men With Metastatic Castration-resistant Prostate Cancer
Brief Title: A Study of Nivolumab or Placebo in Combination With Docetaxel in Men With Advanced Castration-resistant Prostate Cancer
Acronym: CheckMate 7DX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA209-7DX; 2019-002030-36 (EudraCT Number)
Record Dates: First submitted 2019-09-20; First posted 2019-09-23 (Actual); Results first posted 2024-07-22 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Nivolumab; Prednisone; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Nivolumab + docetaxel + prednisone (Experimental)
  Interventions: Biological: Nivolumab; Drug: Prednisone; Drug: Docetaxel
- Arm B: Placebo + docetaxel + prednisone (Placebo Comparator)
  Interventions: Drug: Prednisone; Drug: Docetaxel; Other: Placebo

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: OPDIVO,; BMS-936558-01
  Arms: Arm A: Nivolumab + docetaxel + prednisone
Drug: Prednisone — Specified dose on specified days
Drug: Docetaxel — Specified dose on specified days
Other: Placebo — Specified dose on specified days
  Arms: Arm B: Placebo + docetaxel + prednisone

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of nivolumab with docetaxel in men with advanced castration resistant prostate cancer who have progressed after second-generation hormonal manipulation.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of adenocarcinoma of the prostate without small cell features
* Current evidence of metastatic disease documented by either bone lesions on radionuclide bone scan and/or soft tissue lesions on computerized tomography/magnetic resonance imaging (CT/MRI)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Ongoing androgen deprivation therapy (ADT) with a gonadotropin-releasing hormone (GnRH) analogue or bilateral orchiectomy
* Documented prostate cancer progression per Prostate Cancer Working Group (PCWG3) criteria within 6 months prior to screening
* Chemotherapy-naïve for metastatic castration-resistant prostate cancer (mCRPC), with 1 to 2 prior second generation hormonal therapies in the recurrent non-metastatic setting and/or metastatic setting, and no more than 1 second generation hormonal therapy in the mCRPC setting. Must have progressed during or after second generation hormonal therapy or have documented intolerance to second generation hormonal therapy
* Participants must meet one of the following criteria regarding tissue submission: Sufficient tumor samples from a newly obtained ("fresh") biopsy (obtained during screening); or archival tumor tissue in the form of formalin-fixed paraffin-embedded (FFPE) block or unstained tumor tissue slides. For participants with bone-only disease or inaccessible soft tissue lesions or if the biopsy procedure would pose an unacceptable clinical risk for the participant, submission of tumor tissue obtained from a fresh biopsy is not required.
* Men must agree to follow specific methods of contraception, if applicable

Exclusion Criteria:

* Active brain metastases
* Active, known, or suspected autoimmune disease
* Condition requiring systemic treatment with corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of start of study treatment. Inhaled or topical steroids or adrenal replacement steroid doses are permitted in the absence of active autoimmune disease
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Prior treatment with docetaxel or other chemotherapy for mCRPC. Prior docetaxel for metastatic castration-sensitive prostate cancer is permitted if at least 12 months have elapsed from last dose of docetaxel

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1030 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (293):
- United States (45):
  - Local Institution - 0305, Mobile, Alabama
  - Local Institution - 0012, Anchorage, Alaska
  - Local Institution - 0293, Tucson, Arizona
  - Local Institution - 0269, Jonesboro, Arkansas
  - Local Institution - 0179, Orange, California
  - Local Institution - 0055, Rancho Mirage, California
  - Local Institution - 0260, Redondo Beach, California
  - Local Institution - 0081, Santa Monica, California
  - Local Institution - 0087, Denver, Colorado
  - Local Institution - 0190, West Haven, Connecticut
  - Local Institution - 0366, Washington D.C., District of Columbia
  - Local Institution - 0196, Hollywood, Florida
  - Local Institution - 0397, Jacksonville, Florida
  - Local Institution - 0164, Lakeland, Florida
  - Local Institution - 0181, Orlando, Florida
  - Local Institution - 0285, Pensacola, Florida
  - Local Institution - 0177, Weston, Florida
  - Local Institution - 0117, Atlanta, Georgia
  - Local Institution - 0126, Marietta, Georgia
  - Local Institution - 0382, Thomasville, Georgia
  - Local Institution - 0287, Niles, Illinois
  - Local Institution - 0183, Fort Wayne, Indiana
  - Local Institution - 0302, Louisville, Kentucky
  - Local Institution - 0150, Baltimore, Maryland
  - Local Institution - 0332, Brandywine, Maryland
  - Local Institution - 0299, Omaha, Nebraska
  - Local Institution - 0365, East Brunswick, New Jersey
  - Local Institution - 0139, Florham Park, New Jersey
  - Local Institution - 0300, Albany, New York
  - Local Institution - 0028, Port Jefferson Station, New York
  - Local Institution - 0333, Columbus, Ohio
  - Local Institution - 0180, Allentown, Pennsylvania
  - Local Institution - 0074, Bala-Cynwyd, Pennsylvania
  - Local Institution - 0292, Pittsburgh, Pennsylvania
  - Local Institution - 0233, Charleston, South Carolina
  - Local Institution - 0115, Myrtle Beach, South Carolina
  - Local Institution - 0149, Germantown, Tennessee
  - Local Institution - 0286, Austin, Texas
  - Local Institution - 0303, Dallas, Texas
  - Local Institution - 0284, Houston, Texas
  - Local Institution - 0195, Houston, Texas
  - Local Institution - 0011, San Antonio, Texas
  - The University of Texas Health Science Center at Tyler DBA UT Health East Texas Hope Cancer Center, Tyler, Texas
  - Local Institution - 0110, Seattle, Washington
  - Local Institution - 0289, Spokane, Washington
- Argentina (10):
  - Local Institution - 0129, Mar del Plata, Buenos Aires
  - Local Institution - 0061, Pergamino, Buenos Aires
  - Local Institution - 0153, Parana, Córdoba Province
  - Local Institution - 0393, Río Cuarto, Córdoba Province
  - Local Institution - 0083, Viedma, Río Negro Province
  - Local Institution - 0077, Buenos Aires
  - Local Institution - 0178, Buenos Aires
  - Local Institution - 0185, Buenos Aires
  - Local Institution - 0369, La Rioja
  - Local Institution - 0394, San Juan
- Australia (10):
  - Local Institution - 0152, Gosford, New South Wales
  - Local Institution - 0091, Lismore, New South Wales
  - Local Institution - 0132, Wahroonga, New South Wales
  - Local Institution - 0127, Westmead, New South Wales
  - Local Institution - 0006, South Brisbane, Queensland
  - Local Institution - 0084, Woolloongabba, Queensland
  - Local Institution - 0010, North Adelaide, South Australia
  - Local Institution - 0379, Ballarat, Victoria
  - Local Institution - 0040, Frankston, Victoria
  - Local Institution - 0032, Malvern, Victoria
- Austria (4):
  - Local Institution - 0118, Linz, Upper Austria
  - Local Institution - 0038, Salzburg
  - Local Institution - 0157, Vienna
  - Local Institution - 0131, Vienna
- Belgium (6):
  - Local Institution - 0122, Anderlecht, Brussels Capital
  - Local Institution - 0121, Bruges
  - Local Institution - 0114, Ghent
  - Local Institution - 0162, Ghent
  - Local Institution - 0137, Turnhout
  - Local Institution - 0029, Wilrijk
- Brazil (17):
  - Local Institution - 0097, Belo Horizonte, Minas Gerais
  - Local Institution - 0022, Belo Horizonte, Minas Gerais
  - Local Institution - 0100, Curitiba, Paraná
  - Local Institution - 0082, Curitiba, Paraná
  - Local Institution - 0321, Natal, Rio Grande do Norte
  - Local Institution - 0058, Ijuí, Rio Grande do Sul
  - Local Institution - 0063, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0056, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0057, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0086, Campinas, São Paulo
  - Local Institution - 0059, Santo André, São Paulo
  - Local Institution - 0096, São José do Rio Preto, São Paulo
  - Local Institution - 0189, Rio de Janeiro
  - Local Institution - 0060, Rio de Janeiro
  - Local Institution - 0080, São Paulo
  - Local Institution - 0273, São Paulo
  - Local Institution - 0328, São Paulo
- Canada (3):
  - Local Institution - 0151, Brampton, Ontario
  - Local Institution - 0191, Toronto, Ontario
  - Local Institution - 0143, Montreal, Quebec
- Chile (5):
  - Local Institution - 0027, Viña del Mar, Región de Valparaíso
  - Local Institution - 0026, Santiago, RM
  - Local Institution - 0378, Providencia, Santiago Metropolitan
  - Local Institution - 0025, Santiago, Santiago Metropolitan
  - Local Institution - 0377, Santiago, Santiago Metropolitan
- China (27):
  - Local Institution - 0245, Beijing, Beijing Municipality
  - Local Institution - 0140, Beijing, Beijing Municipality
  - Local Institution - 0254, Beijing, Beijing Municipality
  - Local Institution - 0337, Beijing, Beijing Municipality
  - Local Institution - 0345, Beijing, Beijing Municipality
  - Local Institution - 0312, Beijing, Bei
  - Local Institution - 0256, Fuzhou, Fujian
  - Local Institution - 0319, Guangzhou, Guangdong
  - Local Institution - 0320, Baoding Shi, Hebei
  - Local Institution - 0224, Harbin, Heilongjiang
  - Local Institution - 0314, Henan Sheng, Henan
  - Local Institution - 0275, Zhengzhou, Henan
  - Local Institution - 0313, Wuhan, Hubei
  - Local Institution - 0168, Changsha, Hunan
  - Local Institution - 0165, Nanjing, Jiangsu
  - Local Institution - 0317, Nanjing, Jiangsu
  - Local Institution - 0325, Nanjing, Jiangsu
  - Local Institution - 0347, Nanchang, Jiangxi
  - Local Institution - 0330, Nanchang, Jiangxi
  - Local Institution - 0161, Shenyang, Liaoning
  - Local Institution - 0326, Jinan, Shandong
  - Local Institution - 0155, Shanghai, Shanghai Municipality
  - Local Institution - 0353, Xi'an, Shannxi
  - Local Institution - 0253, Chengdu, Sichuan
  - Local Institution - 0310, Ürümqi, Xinjiang
  - Local Institution - 0316, Hangzhou, Zhejiang
  - Local Institution - 0344, Hangzhou, Zhejiang
- Czechia (6):
  - Local Institution - 0108, Brno
  - Local Institution - 0093, Brno
  - Local Institution - 0049, Olomouc
  - Local Institution - 0088, Ostrava
  - Local Institution - 0050, Prague
  - Local Institution - 0361, Prague
- France (19):
  - Local Institution - 0105, Strasbourg, Alsace
  - Local Institution - 0079, Lille, Nord
  - Local Institution - 0167, Le Mans, Sarthe
  - Local Institution - 0107, Angers
  - Local Institution - 0202, Brest
  - Local Institution - 0398, Dijon
  - Local Institution - 0030, Hyères
  - Local Institution - 0395, Montpellier
  - Local Institution - 0109, Montpellier
  - Local Institution - 0384, Nice
  - Local Institution - 0068, Nîmes
  - Local Institution - 0381, Paris
  - Local Institution - 0106, Paris
  - Local Institution - 0071, Paris
  - Local Institution - 0133, Pierre-Bénite
  - Local Institution - 0399, Reims
  - Local Institution - 0380, Rennes
  - Local Institution - 0387, Strasbourg
  - Local Institution - 0271, Villejuif
- Germany (16):
  - Local Institution - 0023, Nürtingen, Baden-Wurttemberg
  - Local Institution - 0014, Koblenz, Rheinland Pfa
  - Local Institution - 0090, Dresden, Saxony
  - Local Institution - 0089, Bonn
  - Local Institution - 0376, Düsseldorf
  - Local Institution - 0172, Emmendingen
  - Local Institution - 0142, Erlangen
  - Local Institution - 0018, Frankfurt am Main
  - Local Institution - 0064, Hamburg
  - Local Institution - 0069, Hamburg
  - Local Institution - 0389, Heidelberg
  - Local Institution - 0004, Magdeburg
  - Local Institution - 0372, Marburg
  - Local Institution - 0204, München
  - Local Institution - 0036, Münster
  - Local Institution - 0169, Tübingen
- Hong Kong (3):
  - Local Institution - 0145, Hong Kong
  - Local Institution - 0045, Hong Kong
  - Local Institution - 0146, Hong Kong
- Israel (6):
  - Local Institution - 0072, Haifa
  - Local Institution - 0388, Jerusalem
  - Local Institution - 0368, Kfar Saba
  - Local Institution - 0128, Petah Tikva
  - Local Institution - 0135, Ramat Gan
  - Local Institution - 0138, Tel Aviv
- Italy (13):
  - Local Institution - 0099, Benevento
  - Local Institution - 0001, Bergamo
  - Local Institution - 0111, Bologna
  - Local Institution - 0039, Brescia
  - Local Institution - 0053, Cremona
  - Local Institution - 0066, Milan
  - Local Institution - 0120, Napoli
  - Local Institution - 0070, Orbassano
  - Local Institution - 0037, Parma
  - Local Institution - 0199, Pisa
  - Local Institution - 0046, Rome
  - Local Institution - 0385, Rome
  - Local Institution - 0067, Trento
- Japan (24):
  - Local Institution - 0362, Nagoya, Aichi-ken
  - Local Institution - 0340, Akita, Akita
  - Local Institution - 0358, Hirosaki-shi, Aomori
  - Local Institution - 0346, Chiba, Chiba
  - Local Institution - 0339, Sakura-Shi, Chiba
  - Local Institution - 0307, Matsuyama, Ehime
  - Local Institution - 0280, Fukuoka, Fukuoka
  - Local Institution - 0281, Sapporo, Hokkaido
  - Local Institution - 0296, Sapporo, Hokkaido
  - Local Institution - 0283, Yokohama, Kanagawa
  - Local Institution - 0324, Kumamoto, Kumamoto
  - Local Institution - 0342, Kamigyō-ku, Kyoto
  - Local Institution - 0355, Kashihara-shi, Nara
  - Local Institution - 0343, Osaka, Osaka
  - Local Institution - 0323, Ōsaka-sayama, Osaka
  - Local Institution - 0309, Hamamatsu, Shizuoka
  - Local Institution - 0279, Toyama, Toyama
  - Local Institution - 0282, Ube Shi, Yamaguchi
  - Local Institution - 0341, Nagasaki
  - Local Institution - 0327, Niigata
  - Local Institution - 0354, Okayama
  - Local Institution - 0338, Osaka
  - Local Institution - 0308, Tokyo
  - Local Institution - 0278, Wakayama
- Mexico (4):
  - Local Institution - 0017, Mexico City, D.F.
  - Local Institution - 0015, Zapopan, Jalisco
  - Local Institution - 0016, Zapopan, Jalisco
  - Local Institution - 0062, Morelia, Michoacán
- New Zealand (3):
  - Local Institution - 0184, Palmerston North, Manawatu-Wanganui
  - Local Institution - 0101, Hamilton
  - Local Institution - 0102, Tauranga
- Poland (7):
  - Local Institution - 0383, Bydgoszcz
  - Local Institution - 0136, Koszalin
  - Local Institution - 0009, Lodz
  - Local Institution - 0013, Lublin
  - Local Institution - 0065, Poznan
  - Local Institution, Warsaw
  - Local Institution - 0095, Warsaw
- Puerto Rico (2):
  - Local Institution - 0329, Rio Piedras
  - Local Institution - 0359, San Juan
- Romania (6):
  - Local Institution - 0041, Cluj-Napoca, Cluj-Napoca
  - Local Institution - 0042, Bucharest
  - Local Institution - 0043, Cluj-Napoca
  - Local Institution - 0020, Constanța
  - Local Institution - 0052, Craiova
  - Local Institution - 0035, Timișoara
- Russia (10):
  - SBHI Arkhangelsk Region - Arkhangelsk Clinical Oncological Dispensary, Arkhangelsk
  - SAHI Republican Clinical Oncology Dispensary of MoH of RT, Kazan'
  - Clinical Hospital MEDSI in Otradnoye, Krasnogorsk Moscow Region
  - Federal State Budgetary Institution N.N. Blokhin National Medical Research Center of Oncology of the, Moscow
  - Sechenov University, Moscow
  - P.A. Herzen Moscow Oncology Research Institute, Moscow
  - FSBI National Medical Research Radiology Center NMRRC - A. Tsyb Medical Radiological Research Centre, Obninsk
  - Budgetary Healthcare Institution of Omsk Region &quot,Clinical Oncological Dispensary&quot,, Omsk
  - Andros Clinic LLC, Saint Petersburg
  - Russian Scientific Centre of Radiology and Surgical Technologies n.a. acad. M.A., Saint Petersburg
- Singapore (3):
  - Local Institution - 0116, Singapore
  - Local Institution - 0005, Singapore
  - Local Institution - 0170, Singapore
- South Korea (12):
  - Local Institution - 0297, Jung-gu, Daejeon
  - Local Institution - 0186, Songnam-si, Gyeonggi-do
  - Local Institution - 0391, Daegu
  - Local Institution - 0298, Incheon
  - Local Institution - 0375, Jeollanam-do
  - Local Institution - 0374, Seodaemun-Gu
  - Local Institution - 0370, Seoul
  - Local Institution - 0171, Seoul
  - Local Institution - 0193, Seoul
  - Local Institution - 0187, Seoul
  - Local Institution - 0373, Seoul
  - Local Institution - 0158, Yangsan
- Spain (13):
  - Local Institution - 0141, Manresa, Barcelona
  - Local Institution - 0073, Barcelona
  - Local Institution - 0123, Barcelona
  - Local Institution - 0360, Córdoba
  - Local Institution - 0044, Girona
  - Local Institution - 0034, Lugo
  - Local Institution - 0076, Madrid
  - Local Institution - 0024, Madrid
  - Local Institution - 0003, Madrid
  - Local Institution - 0031, Madrid
  - Local Institution - 0364, Madrid
  - Local Institution - 0124, Sabadell (Barcelona)
  - Local Institution - 0363, Seville
- Taiwan (6):
  - Local Institution - 0192, Niaosng, Kaohsiung
  - Local Institution - 0194, Taichung
  - Local Institution - 0371, Taichung
  - Local Institution - 0386, Tainan
  - Local Institution - 0175, Taipei
  - Local Institution - 0188, Taipei
- Turkey (Türkiye) (6):
  - Local Institution - 0094, Adana
  - Local Institution - 0119, Ankara
  - Local Institution - 0130, Ankara
  - Local Institution - 0113, Istanbul
  - Local Institution - 0104, Izmir
  - Local Institution - 0112, Malatya
- United Kingdom (7):
  - Local Institution - 0173, London, Greater London
  - Local Institution - 0098, Manchester, Lancashire
  - Local Institution - 0008, Northwood, Middlesex
  - Local Institution - 0051, Nottingham, Nottinghamshire
  - Local Institution - 0265, Oxford, Oxfordshire
  - Local Institution - 0048, Guildford, Surrey
  - Local Institution - 0154, London

REFERENCES:
- [Derived] Fizazi K, Saad F, Alonso-Gordoa T, Zurawski B, Barthelemy P, Voog E, Cutuli HJ, Buchler T, Ye D, Castellano D, Kwiatkowski M, Arslan C, Richardet M, Alifrangis C, Goh JC, Vianna K, Han W, Hatano K, Todenhofer T, Retz M, Srivastava A, Jin C, Gupta S, Trandafirescu G, Campos A, Lee CW, van Kooten Losio M, Subudhi SK. Nivolumab plus docetaxel versus placebo plus docetaxel for androgen receptor pathway inhibitor-pretreated and chemotherapy-naive metastatic castration-resistant prostate cancer (CheckMate 7DX): a double-blind, randomised, phase 3 trial. Lancet Oncol. 2026 Jan;27(1):68-78. doi: 10.1016/S1470-2045(25)00566-2. PMID 41449150
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab + Docetaxel + Prednisone: Participants with metastatic castration resistant prostate cancer (mCRPC) who are chemotherapy-naïve for mCRPC and have received at least 1 but no more than 2 second-generation hormonal manipulations received Docetaxel 75 milligram per meter square (mg/m^2) intravenous (IV) once in a week (Q3W) + Prednisone 5 milligram (mg) orally (PO) twice a day (BID) + Nivolumab 360 mg IV Q3W for maximum 10 cycles, followed by Nivolumab 480 mg IV once in four weeks (Q4W) until disease progression or unacceptable toxicity or maximum of 2 years from the date of first dose or withdraw of consent.
- Placebo + Docetaxel + Prednisone: Participants with metastatic castration resistant prostate cancer (mCRPC) who are chemotherapy-naïve for mCRPC and have received at least 1 but no more than 2 second-generation hormonal manipulations received Docetaxel 75 mg/m^2 IV Q3W + Prednisone 5 mg PO BID + Placebo IV Q3W for maximum 10 cycles, followed by Placebo IV Q4W until disease progression or unacceptable toxicity or maximum of 2 years from the date of first dose or withdraw of consent.
Period: Pre-Treatment Period
Arm/Group | Nivolumab + Docetaxel + Prednisone | Placebo + Docetaxel + Prednisone
Started | 514 | 516
Completed | 510 | 510
Not Completed | 4 | 6
Not completed — Not Reported | 0 | 4
Not completed — Subject no longer meets study criteria | 1 | 1
Not completed — Poor/Non-compliance | 1 | 0
Not completed — Participant withdrew consent | 2 | 0
Not completed — Participant request to discontinue study treatment | 0 | 1
Period: Treatment Period
Arm/Group | Nivolumab + Docetaxel + Prednisone | Placebo + Docetaxel + Prednisone
Started | 510 | 510
Completed | 19 | 11
Not Completed | 491 | 499
Not completed — Ongoing Treatment | 1 | 0
Not completed — Other Reason | 26 | 37
Not completed — Completed treatment as per protocol | 1 | 2
Not completed — Maximum clinical benefit | 3 | 0
Not completed — Adverse event unrelated to study drug | 13 | 12
Not completed — Study drug toxicity | 67 | 28
Not completed — Disease Progression | 284 | 327
Not completed — Administrative reasons by sponsor | 16 | 30
Not completed — Poor/Non-Compliance | 1 | 0
Not completed — Lost to Follow-up | 2 | 2
Not completed — Death | 16 | 11
Not completed — Participant withdrew consent | 10 | 10
Not completed — Participant request to discontinue study treatment | 33 | 32
Not completed — Adverse Event | 14 | 6
Not completed — Lack of Efficacy | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab + Docetaxel + Prednisone | Placebo + Docetaxel + Prednisone | Total
Number analyzed (Participants) | 514 | 516 | 1030
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (7.5) | 69.6 (8.1) | 69.2 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 514 | 515 | 1029
Race/Ethnicity, Customized [Number; unit: participants]
  White | 333 | 329 | 662
  Black or African American | 20 | 15 | 35
  Asian | 35 | 45 | 80
  Native Hawaiian or other pacific islander | 1 | 0 | 1
  Chinese | 40 | 38 | 78
  Japanese | 33 | 45 | 78
  Asian other | 1 | 0 | 1
  Other | 30 | 27 | 57
  Not Reported | 19 | 16 | 35
  Asian Indian | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Progressive Free Survival (rPFS) Assessed by Blinded Independent Central Review (BICR) Per Prostate Cancer Working Group 3 (PCWG3)
Description: rPFS for randomized participants is the time between randomization and the first date of documented progression or death due to any cause, whichever occurs first. The rPFS was censored at the last radiographic tumor assessment up to the start of subsequent cancer therapy for those without progression or death. It was also censored at the date of last radiographic tumor assessment prior to the missed tumor assessments for participants who had progressive disease (PD) or death immediately after more than one consecutive missed tumor assessments. Radiographic progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeter (mm). The appearance of one or more new lesions is also considered progression.
Time Frame: from randomization to the first date of documented progression or death due to any cause, whichever occurs first (up to approximately 31 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab + Docetaxel + Prednisone | Placebo + Docetaxel + Prednisone
Number analyzed (Participants) | 514 | 516
months | 9.43 [8.48 to 10.32] | 8.74 [8.38 to 9.99]
Statistical Analysis 1: Comparison: Nivolumab + Docetaxel + Prednisone vs Placebo + Docetaxel + Prednisone; Test type: Superiority; p = 0.5901, Log Rank — Boundary for statistical significance p-value < 0.01; Stratification factor is visceral disease (YES vs NO) as entered in the IRT; Cox Proportional Hazard = 0.96, 99% CI 2-sided [0.77 to 1.19]

2. Primary Outcome: Overall Survival (OS)
Description: OS for all randomized participants is the time between randomization and the date of death from any cause. For participants who are alive, their survival time was censored at the last date that they were known to be alive. OS was censored for participants at the date of randomization if they had no follow-up.
Time Frame: From randomization to the date of death from any cause (Up to approximately 31 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab + Docetaxel + Prednisone | Placebo + Docetaxel + Prednisone
Number analyzed (Participants) | 514 | 516
months | 18.73 [16.95 to 21.03] | 18.92 [17.31 to 22.01]
Statistical Analysis 1: Comparison: Nivolumab + Docetaxel + Prednisone vs Placebo + Docetaxel + Prednisone; Test type: Superiority; p = 0.3572, Log Rank — Boundary for statistical significance p-value < 0.0059. Additional accuracy for p-value: 0.005866; Cox Proportional Hazard = 1.09, 99.41% CI 2-sided [0.84 to 1.43] — Stratification factor is visceral disease (YES vs NO) as entered in the IRT

3. Secondary Outcome: Objective Response Rate (ORR) Assessed by Blinded Independent Central Review (BICR) Per Prostate Cancer Working Group (PCWG3)
Description: Objective Response Rate per PCWG3 (ORR-PCWG3) is the percentage of participants who have a confirmed complete or partial best overall response (BOR) per PCWG3 among randomized participants who have measurable disease at baseline. Complete Response (CR) is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial Response (PR) is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Baseline was defined as evaluations or events that occur before the date and time of the first dose of study treatment or evaluations on the same date and time of the first dose of study treatment were also considered as baseline evaluations.
Time Frame: From date of randomization to the date of objectively documented progression per PCWG3 or the date of subsequent systemic cancer therapy, whichever occurs first (Up to approximately 52 months)
Population: All response evaluable participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nivolumab + Docetaxel + Prednisone | Placebo + Docetaxel + Prednisone
Number analyzed (Participants) | 216 | 204
percentage of participants | 27.3 [21.5 to 33.8] | 23.5 [17.9 to 30.0]
Statistical Analysis 1: Comparison: Nivolumab + Docetaxel + Prednisone vs Placebo + Docetaxel + Prednisone; Test type: Superiority; Adjusted Difference = 3.8, 95% CI 2-sided [-4.5 to 12.1] — Strata adjusted difference in objective response rate based on DerSimonian and Laird method. Stratified by visceral disease (YES vs NO) as entered in the IRT

4. Secondary Outcome: Time to Response (TTR) Assessed by Blinded Independent Central Review (BICR) Per Prostate Cancer Working Group (PCWG3)
Description: Time to Response per PCWG3 (TTR-PCWG3) is the time from randomization to the date of the first documented CR or PR per PCWG3, as determined by BICR. Complete Response (CR) is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial Response (PR) is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From randomization to the date of the first documented CR or PR (Up to approximately 52 months)
Population: All Confirmed Responders (PR + CR)
Measure: Median (Full Range); unit: months
Arm/Group | Nivolumab + Docetaxel + Prednisone | Placebo + Docetaxel + Prednisone
Number analyzed (Participants) | 59 | 48
months | 2.17 [1.4 to 7.8] | 2.20 [1.7 to 8.2]

5. Secondary Outcome: Duration of Response Assessed by Blinded Independent Central Review (BICR) Per Prostate Cancer Working Group (PCWG3)
Description: Duration of Response per PCWG3 (DOR-PCWG3) is time between the date of first response (CR/PR per PCWG3) to the date of first documented radiographic progression per PCWG3,as determined by BICR, or death due to any cause whichever occurs first. Complete Response (CR) is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial Response (PR) is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Radiographic progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeter (mm). The appearance of one or more new lesions is also considered progression.
Time Frame: From randomization date to the date of first documented radiographic progression or death due to any cause whichever occurs first (Up to approximately 52 months)
Population: All Confirmed Responders (PR + CR)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab + Docetaxel + Prednisone | Placebo + Docetaxel + Prednisone
Number analyzed (Participants) | 59 | 48
months | 8.31 [6.18 to 10.15] | 8.11 [6.34 to 8.74]

6. Secondary Outcome: Prostate-specific Antigen (PSA) Response Rate (PSA-RR)
Description: PSA Response Rate (PSA-RR) is the percentage of randomized participants with a 50% or greater decrease in PSA from baseline to the lowest post-baseline PSA result. A second consecutive value obtained 3 or more weeks later is required to confirm the PSA response. Baseline was defined as valuations or events that occur before the date and time of the first dose of study treatment or evaluations on the same date and time of the first dose of study treatment were also considered as baseline evaluations.
Time Frame: Up to approximately 52 months
Population: All randomized participants with baseline and at least one post-baseline PSA assessments
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nivolumab + Docetaxel + Prednisone | Placebo + Docetaxel + Prednisone
Number analyzed (Participants) | 498 | 503
percentage of participants | 42.4 [38.0 to 46.8] | 41.6 [37.2 to 46.0]
Statistical Analysis 1: Comparison: Nivolumab + Docetaxel + Prednisone vs Placebo + Docetaxel + Prednisone; Test type: Superiority; Percentage Difference = 0.9, 95% CI 2-sided [-5.2 to 7.0] — [estimate comment as in outcome 3, analysis 1]

7. Secondary Outcome: Time to PSA Progression (TTP-PSA)
Description: Time to PSA Progression (TTP-PSA) is the time between randomization to the date of PSA progression per PCWG3 in randomized participants. PSA Progression: For participants with an initial PSA decline from baseline, the date of PSA progression is the date that an increase of 25% or more and an absolute increase of 2 ng/mL or more from the nadir are documented and confirmed by a second consecutive PSA value at least 3 weeks later. For participants with no PSA decline from baseline, the date of PSA progression is date that an increase of 25% or more and an absolute increase of 2 ng/mL or more from baseline are documented at or beyond Week 13. Baseline was defined as valuations or events that occur before the date and time of the first dose of study treatment or evaluations on the same date and time of the first dose of study treatment were also considered as baseline evaluations. Censored at date of last PSA evaluation on/prior to start of subsequent cancer therapy.
Time Frame: from randomization to the date of PSA Progression (Up to approximately 31 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab + Docetaxel + Prednisone | Placebo + Docetaxel + Prednisone
Number analyzed (Participants) | 514 | 516
months | 6.28 [5.82 to 6.97] | 6.21 [5.65 to 6.77]
Statistical Analysis 1: Comparison: Nivolumab + Docetaxel + Prednisone vs Placebo + Docetaxel + Prednisone; Test type: Superiority; Cox Proportional Hazard = 1.00, 95% CI 2-sided [0.86 to 1.16] — Stratification factor is visceral disease (YES vs NO) as entered in the IRT

8. Secondary Outcome: Number of Participants With Adverse Events
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: From first dose and 30 days after last dose of study therapy (Up to approximately 25 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Docetaxel + Prednisone | Placebo + Docetaxel + Prednisone
Number analyzed (Participants) | 510 | 510
Participants | 501 | 503

9. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose results in death or Is life-threatening or requires inpatient hospitalization or causes prolongation of existing hospitalization or results in persistent or significant disability/incapacity or is a congenital anomaly/birth defect.
Time Frame: From first dose and 30 days after last dose of study therapy (Up to approximately 25 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Docetaxel + Prednisone | Placebo + Docetaxel + Prednisone
Number analyzed (Participants) | 510 | 510
Participants | 223 | 192

10. Secondary Outcome: Number of Participants With Adverse Events Leading to Discontinuation
Description: as for outcome 8
Time Frame: From first dose and 30 days after last dose of study therapy (Up to approximately 25 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Docetaxel + Prednisone | Placebo + Docetaxel + Prednisone
Number analyzed (Participants) | 510 | 510
Participants | 148 | 101

11. Secondary Outcome: Number of Participants With Endocrine Immune-Mediated Adverse Events
Description: Immune-mediated adverse events are AEs consistent with an immune-mediated mechanism or immune-mediated component for which non-inflammatory etiologies (eg, infection or tumor progression) have been ruled out. IMAEs can include events with an alternate etiology which were exacerbated by the induction of autoimmunity. An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: From first dose and 100 days after last dose of study therapy (Up to approximately 13 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Docetaxel + Prednisone | Placebo + Docetaxel + Prednisone
Number analyzed (Participants) | 510 | 510
Participants
  Adrenal insufficiency | 7 | 4
  Hypothyroidism | 27 | 11
  Thyroiditis | 1 | 0
  Diabetes mellitus | 1 | 2
  Diabetic ketoacidosis | 1 | 0
  Type 1 diabetes mellitus | 1 | 0
  Hyperthyroidism | 20 | 11
  Immune-mediated hypophysitis | 1 | 0
  Hypopituitarism | 0 | 1

12. Secondary Outcome: Number of Participants With Non-Endocrine Immune-Mediated Adverse Events
Description: as for outcome 11
Time Frame: From first dose and 100 days after last dose of study therapy (Up to approximately 13 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Docetaxel + Prednisone | Placebo + Docetaxel + Prednisone
Number analyzed (Participants) | 510 | 510
Participants
  Pneumonitis | 15 | 2
  Interstitial lung disease | 5 | 1
  Immune-mediated lung disease | 1 | 0
  Diarrhoea | 8 | 2
  Colitis | 4 | 0
  Enterocolitis | 1 | 0
  Alanine aminotransferase increased | 5 | 0
  Aspartate aminotransferase increased | 3 | 0
  Hypertransaminasaemia | 3 | 0
  Autoimmune hepatitis | 2 | 0
  Immune-mediated hepatitis | 2 | 0
  Blood bilirubin increased | 1 | 0
  Cholangitis | 1 | 0
  Blood creatinine increased | 1 | 0
  Acute kidney injury | 0 | 1
  Immune-mediated nephritis | 0 | 1
  Rash | 14 | 7
  Rash maculo-papular | 3 | 0
  Rash pustular | 2 | 0
  Dermatitis | 1 | 1
  Dermatitis acneiform | 1 | 0
  Drug eruption | 1 | 0
  Pemphigoid | 1 | 0
  Erythema multiforme | 0 | 1
  Immune-mediated dermatitis | 0 | 1
  Rash macular | 0 | 1
  Infusion related reaction | 3 | 3
  Hypersensitivity | 0 | 1
  Infusion related hypersensitivity reaction | 0 | 1

13. Secondary Outcome: Number of Participants With Select Adverse Events
Description: as for outcome 8
Time Frame: From first dose and 30 days after last dose of study therapy (Up to approximately 25 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Docetaxel + Prednisone | Placebo + Docetaxel + Prednisone
Number analyzed (Participants) | 510 | 510
Participants
  Diarrhoea | 176 | 159
  Colitis | 7 | 2
  Enterocolitis | 2 | 1
  Frequent bowel movements | 0 | 1
  Alanine aminotransferase increased | 36 | 14
  Aspartate aminotransferase increased | 26 | 15
  Blood alkaline phosphatase increased | 23 | 22
  Blood bilirubin increased | 8 | 4
  Gamma-glutamyltransferase increased | 5 | 3
  Hepatic cytolysis | 4 | 1
  Transaminases increased | 4 | 1
  Autoimmune hepatitis | 2 | 0
  Cholangitis | 2 | 0
  Hyperbilirubinaemia | 2 | 2
  Hypertransaminasaemia | 2 | 0
  Hepatic enzyme increased | 1 | 2
  Hepatitis | 1 | 0
  Immune-mediated hepatitis | 1 | 0
  Liver injury | 1 | 0
  Liver disorder | 0 | 1
  Pneumonitis | 26 | 6
  Interstitial lung disease | 7 | 4
  Acute respiratory failure | 1 | 0
  Immune-mediated lung disease | 1 | 0
  Lung infiltration | 1 | 0
  Idiopathic interstitial pneumonia | 0 | 1
  Blood creatinine increased | 22 | 7
  Acute kidney injury | 7 | 9
  Renal failure | 3 | 5
  Blood urea increased | 2 | 2
  Immune-mediated nephritis | 0 | 1
  Rash | 51 | 34
  Pruritus | 47 | 20
  Eczema | 10 | 3
  Rash maculo-papular | 11 | 6
  Dermatitis | 6 | 4
  Palmar-plantar erythrodysaesthesia syndrome | 5 | 22
  Urticaria | 5 | 3
  Erythema | 4 | 11
  Psoriasis | 4 | 3
  Skin exfoliation | 4 | 2
  Dermatitis acneiform | 3 | 1
  Rash macular | 3 | 2
  Dermatitis allergic | 2 | 0
  Rash erythematous | 2 | 2
  Rash pustular | 3 | 0
  Vitiligo | 2 | 1
  Blister | 1 | 0
  Dermatitis atopic | 1 | 2
  Dermatitis exfoliative | 1 | 0
  Drug eruption | 1 | 0
  Erythema multiforme | 1 | 1
  Exfoliative rash | 1 | 0
  Pemphigoid | 1 | 0
  Photosensitivity reaction | 1 | 0
  Rash papular | 1 | 1
  Rash pruritic | 1 | 0
  Immune-mediated dermatitis | 0 | 1
  Infusion related reaction | 22 | 27
  Hypersensitivity | 6 | 4
  Anaphylactic reaction | 1 | 0
  Anaphylactic shock | 1 | 0
  Bronchospasm | 0 | 1
  Infusion related hypersensitivity reaction | 0 | 3

14. Secondary Outcome: Number of Participants Who Died
Time Frame: Up to approximately 52 months
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Docetaxel + Prednisone | Placebo + Docetaxel + Prednisone
Number analyzed (Participants) | 510 | 510
Participants | 258 | 227

15. Secondary Outcome: Number of Participants With Worst Common Terminology Criteria (CTC) Grade Laboratory Test Grade Change From Baseline
Description: The severity of laboratory test results were graded based upon the participants symptoms according to the Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0); Hematology parameters were evaluated for severity according to the following scale: Grade 0 is defined as absence of an AE or within normal limits; Grade 1 = Mild - transient or mild discomfort; no medical intervention required; Grade 2 = Moderate - mild to moderate limitation in activity; Grade 3 = Severe; Grade 4 = Life threatening. Number of participants with worst grade change results to Grade 3 or Grade 4 laboratory test results is presented. E.g., the row title HEMOGLOBIN Grade 0 to Grade 3, Grade 0 is baseline and Grade 3 is post baseline.
Time Frame: From first dose and 30 days after last dose of study therapy (Up to approximately 25 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Docetaxel + Prednisone | Placebo + Docetaxel + Prednisone
Number analyzed (Participants) | 510 | 510
Participants
  HEMOGLOBIN Grade 0 to Grade 3 | 5 | 3
  HEMOGLOBIN Grade 0 to Grade 4 | NA — Per Anemia criteria in CTC version 5.0 there is no grade 4 for hemoglobin | NA — Per Anemia criteria in CTC version 5.0 there is no grade 4 for hemoglobin
  HEMOGLOBIN Grade 1 to Grade 3 | 20 | 16
  HEMOGLOBIN Grade 1 to Grade 4 | NA — Per Anemia criteria in CTC version 5.0 there is no grade 4 for hemoglobin | NA — Per Anemia criteria in CTC version 5.0 there is no grade 4 for hemoglobin
  HEMOGLOBIN Grade 2 to Grade 3 | 11 | 11
  HEMOGLOBIN Grade 2 to Grade 4 | NA — Per Anemia criteria in CTC version 5.0 there is no grade 4 for hemoglobin | NA — Per Anemia criteria in CTC version 5.0 there is no grade 4 for hemoglobin
  HEMOGLOBIN Grade 3 to Grade 3 | 0 | 0
  HEMOGLOBIN Grade 3 to Grade 4 | NA — Per Anemia criteria in CTC version 5.0 there is no grade 4 for hemoglobin | NA — Per Anemia criteria in CTC version 5.0 there is no grade 4 for hemoglobin
  PLATELET COUNT Grade 0 to Grade 3 | 2 | 3
  PLATELET COUNT Grade 0 to Grade 4 | 0 | 1
  PLATELET COUNT Grade 1 to Grade 3 | 2 | 1
  PLATELET COUNT Grade 1 to Grade 4 | 1 | 1
  PLATELET COUNT Grade 2 to Grade 3 | 0 | 0
  PLATELET COUNT Grade 2 to Grade 4 | 0 | 0
  PLATELET COUNT Grade 3 to Grade 3 | 0 | 0
  PLATELET COUNT Grade 3 to Grade 4 | 0 | 0
  PLATELET COUNT Grade 4 to Grade 3 | 0 | 0
  PLATELET COUNT Grade 4 to Grade 4 | 0 | 0
  LEUKOCYTES Grade 0 to Grade 3 | 30 | 28
  LEUKOCYTES Grade 0 to Grade 4 | 11 | 13
  LEUKOCYTES Grade 1 to Grade 3 | 5 | 3
  LEUKOCYTES Grade 1 to Grade 4 | 1 | 1
  LEUKOCYTES Grade 2 to Grade 3 | 0 | 1
  LEUKOCYTES Grade 2 to Grade 4 | 0 | 0
  LEUKOCYTES Grade 3 to Grade 3 | 0 | 0
  LEUKOCYTES Grade 3 to Grade 4 | 0 | 0
  LEUKOCYTES Grade 4 to Grade 3 | 0 | 0
  LEUKOCYTES Grade 4 to Grade 4 | 0 | 0
  LYMPHOCYTES Grade 0 to Grade 3 | 22 | 17
  LYMPHOCYTES Grade 0 to Grade 4 | 1 | 1
  LYMPHOCYTES Grade 1 to Grade 3 | 24 | 22
  LYMPHOCYTES Grade 1 to Grade 4 | 3 | 1
  LYMPHOCYTES Grade 2 to Grade 3 | 19 | 30
  LYMPHOCYTES Grade 2 to Grade 4 | 2 | 2
  LYMPHOCYTES Grade 3 to Grade 3 | 10 | 19
  LYMPHOCYTES Grade 3 to Grade 4 | 2 | 4
  LYMPHOCYTES Grade 4 to Grade 3 | 0 | 0
  LYMPHOCYTES Grade 4 to Grade 4 | 0 | 0
  ANC Grade 0 to Grade 3 | 18 | 16
  ANC Grade 0 to Grade 4 | 44 | 39
  ANC Grade 1 to Grade 3 | 0 | 0
  ANC Grade 1 to Grade 4 | 0 | 1
  ANC Grade 2 to Grade 3 | 0 | 1
  ANC Grade 2 to Grade 4 | 0 | 1
  ANC Grade 3 to Grade 3 | 0 | 0
  ANC Grade 3 to Grade 4 | 0 | 0
  ANC Grade 4 to Grade 3 | 0 | 0
  ANC Grade 4 to Grade 4 | 0 | 0
  ALP Grade 0 to Grade 3 | 5 | 1
  ALP Grade 0 to Grade 4 | 0 | 0
  ALP Grade 1 to Grade 3 | 1 | 1
  ALP Grade 1 to Grade 4 | 0 | 0
  ALP Grade 2 to Grade 3 | 0 | 0
  ALP Grade 2 to Grade 4 | 0 | 0
  ALP Grade 3 to Grade 4 | 0 | 0
  ALP Grade 4 to Grade 3 | 0 | 0
  ALP Grade 4 to Grade 4 | 0 | 0
  AMT Grade 0 to Grade 3 | 6 | 0
  AMT Grade 0 to Grade 4 | 1 | 0
  AMT Grade 1 to Grade 3 | 1 | 2
  AMT Grade 1 to Grade 4 | 1 | 1
  AMT Grade 2 to Grade 3 | 0 | 0
  AMT Grade 2 to Grade 4 | 0 | 0
  AMT Grade 3 to Grade 3 | 0 | 0
  AMT Grade 3 to Grade 4 | 0 | 0
  AMT Grade 4 to Grade 3 | 0 | 0
  AMT Grade 4 to Grade 4 | 0 | 0
  ALT Grade 0 to Grade 3 | 7 | 2
  ALT Grade 0 to Grade 4 | 3 | 0
  ALT Grade 1 to Grade 3 | 0 | 0
  ALT Grade 1 to Grade 4 | 0 | 0
  ALT Grade 2 to Grade 3 | 0 | 0
  ALT Grade 3 to Grade 3 | 0 | 0
  ALT Grade 4 to Grade 3 | 0 | 0
  ALT Grade 4 to Grade 4 | 0 | 0
  BILIRUBIN Grade 0 to Grade 3 | 2 | 1
  BILIRUBIN Grade 0 to Grade 4 | 1 | 0
  BILIRUBIN Grade 1 to Grade 3 | 0 | 0
  BILIRUBIN Grade 1 to Grade 4 | 0 | 0
  BILIRUBIN Grade 2 to Grade 3 | 0 | 0
  BILIRUBIN Grade 2 to Grade 4 | 0 | 0
  BILIRUBIN Grade 3 to Grade 3 | 0 | 0
  BILIRUBIN Grade 3 to Grade 4 | 0 | 0
  BILIRUBIN Grade 4 to Grade 3 | 0 | 0
  BILIRUBIN Grade 4 to Grade 4 | 0 | 0
  CREATININE Grade 0 to Grade 3 | 4 | 4
  CREATININE Grade 0 to Grade 4 | 0 | 0
  CREATININE Grade 1 to Grade 3 | 1 | 0
  CREATININE Grade 1 to Grade 4 | 1 | 0
  CREATININE Grade 2 to Grade 3 | 0 | 1
  CREATININE Grade 2 to Grade 4 | 1 | 0
  CREATININE Grade 3 to Grade 3 | 0 | 0
  CREATININE Grade 3 to Grade 4 | 0 | 0
  CREATININE Grade 4 to Grade 3 | 0 | 0
  CREATININE Grade 4 to Grade 4 | 0 | 0
  HYPERNATREMIA Grade 0 to Grade 3 | 0 | 0
  HYPERNATREMIA Grade 0 to Grade 4 | 0 | 0
  HYPERNATREMIA Grade 1 to Grade 3 | 0 | 0
  HYPERNATREMIA Grade 1 to Grade 4 | 0 | 0
  HYPERNATREMIA Grade 2 to Grade 3 | 0 | 0
  HYPERNATREMIA Grade 2 to Grade 4 | 0 | 0
  HYPERNATREMIA Grade 3 to Grade 3 | 0 | 0
  HYPERNATREMIA Grade 3 to Grade 4 | 0 | 0
  HYPERNATREMIA Grade 4 to Grade 3 | 0 | 0
  HYPERNATREMIA Grade 4 to Grade 4 | 0 | 0
  HYPONATREMIA Grade 0 to Grade 3 | 5 | 4
  HYPONATREMIA Grade 0 to Grade 4 | 0 | 1
  HYPONATREMIA Grade 1 to Grade 3 | 0 | 0
  HYPONATREMIA Grade 1 to Grade 4 | 0 | 1
  HYPONATREMIA Grade 2 to Grade 3 | 0 | 0
  HYPONATREMIA Grade 2 to Grade 4 | 0 | 0
  HYPONATREMIA Grade 3 to Grade 3 | 0 | 0
  HYPONATREMIA Grade 3 to Grade 4 | 0 | 0
  HYPONATREMIA Grade 4 to Grade 3 | 0 | 0
  HYPONATREMIA Grade 4 to Grade 4 | 0 | 0
  HYPERKALEMIA Grade 0 to Grade 3 | 8 | 1
  HYPERKALEMIA Grade 0 to Grade 4 | 2 | 1
  HYPERKALEMIA Grade 1 to Grade 3 | 2 | 0
  HYPERKALEMIA Grade 1 to Grade 4 | 0 | 1
  HYPERKALEMIA Grade 2 to Grade 3 | 1 | 0
  HYPERKALEMIA Grade 2 to Grade 4 | 0 | 0
  HYPERKALEMIA Grade 3 to Grade 3 | 0 | 0
  HYPERKALEMIA Grade 3 to Grade 4 | 0 | 0
  HYPERKALEMIA Grade 4 to Grade 3 | 0 | 0
  HYPERKALEMIA Grade 4 to Grade 4 | 0 | 0
  HYPOKALEMIA Grade 0 to Grade 3 | 7 | 8
  HYPOKALEMIA Grade 0 to Grade 4 | 1 | 0
  HYPOKALEMIA Grade 1 to Grade 3 | 3 | 1
  HYPOKALEMIA Grade 1 to Grade 4 | 0 | 0
  HYPOKALEMIA Grade 2 to Grade 3 | 0 | 0
  HYPOKALEMIA Grade 2 to Grade 4 | 0 | 0
  HYPOKALEMIA Grade 3 to Grade 3 | 0 | 0
  HYPOKALEMIA Grade 3 to Grade 4 | 0 | 0
  HYPOKALEMIA Grade 4 to Grade 3 | 0 | 0
  HYPOKALEMIA Grade 4 to Grade 4 | 0 | 0
  HYPERCALCEMIA Grade 0 to Grade 3 | 0 | 0
  HYPERCALCEMIA Grade 0 to Grade 4 | 0 | 0
  HYPERCALCEMIA Grade 1 to Grade 3 | 0 | 0
  HYPERCALCEMIA Grade 1 to Grade 4 | 1 | 0
  HYPERCALCEMIA Grade 2 to Grade 3 | 0 | 0
  HYPERCALCEMIA Grade 2 to Grade 4 | 0 | 0
  HYPERCALCEMIA Grade 3 to Grade 3 | 0 | 0
  HYPERCALCEMIA Grade 3 to Grade 4 | 0 | 0
  HYPERCALCEMIA Grade 4 to Grade 3 | 0 | 0
  HYPERCALCEMIA Grade 4 to Grade 4 | 0 | 0
  HYPOCALCEMIA Grade 0 to Grade 3 | 6 | 4
  HYPOCALCEMIA Grade 0 to Grade 4 | 1 | 0
  HYPOCALCEMIA Grade 1 to Grade 3 | 1 | 2
  HYPOCALCEMIA Grade 1 to Grade 4 | 0 | 0
  HYPOCALCEMIA Grade 2 to Grade 3 | 3 | 0
  HYPOCALCEMIA Grade 2 to Grade 4 | 3 | 0
  HYPOCALCEMIA Grade 3 to Grade 3 | 0 | 0
  HYPOCALCEMIA Grade 3 to Grade 4 | 0 | 0
  HYPOCALCEMIA Grade 4 to Grade 3 | 0 | 0
  HYPOCALCEMIA Grade 4 to Grade 4 | 0 | 0
  HYPERMAGNESEMIA Grade 0 to Grade 3 | 4 | 3
  HYPERMAGNESEMIA Grade 0 to Grade 4 | 0 | 0
  HYPERMAGNESEMIA Grade 1 to Grade 3 | 1 | 0
  HYPERMAGNESEMIA Grade 1 to Grade 4 | 0 | 0
  HYPERMAGNESEMIA Grade 2 to Grade 3 | 0 | 0
  HYPERMAGNESEMIA Grade 2 to Grade 4 | 0 | 0
  HYPERMAGNESEMIA Grade 3 to Grade 3 | 1 | 0
  HYPERMAGNESEMIA Grade 3 to Grade 4 | 0 | 0
  HYPERMAGNESEMIA Grade 4 to Grade 3 | 0 | 0
  HYPERMAGNESEMIA Grade 4 to Grade 4 | 0 | 0
  HYPOMAGNESEMIA Grade 0 to Grade 3 | 0 | 0
  HYPOMAGNESEMIA Grade 0 to Grade 4 | 0 | 0
  HYPOMAGNESEMIA Grade 1 to Grade 3 | 0 | 0
  HYPOMAGNESEMIA Grade 1 to Grade 4 | 0 | 0
  HYPOMAGNESEMIA Grade 2 to Grade 3 | 0 | 0
  HYPOMAGNESEMIA Grade 2 to Grade 4 | 0 | 0
  HYPOMAGNESEMIA Grade 3 to Grade 3 | 0 | 0
  HYPOMAGNESEMIA Grade 3 to Grade 4 | 0 | 0
  HYPOMAGNESEMIA Grade 4 to Grade 3 | 0 | 0
  HYPOMAGNESEMIA Grade 4 to Grade 4 | 0 | 0
  HYPOGLYCEMIA Grade 0 to Grade 3 | 1 | 1
  HYPOGLYCEMIA Grade 0 to Grade 4 | 1 | 0
  HYPOGLYCEMIA Grade 1 to Grade 3 | 0 | 0
  HYPOGLYCEMIA Grade 1 to Grade 4 | 0 | 0
  HYPOGLYCEMIA Grade 2 to Grade 3 | 0 | 0
  HYPOGLYCEMIA Grade 2 to Grade 4 | 0 | 0
  HYPOGLYCEMIA Grade 3 to Grade 3 | 0 | 0
  HYPOGLYCEMIA Grade 3 to Grade 4 | 0 | 0
  HYPOGLYCEMIA Grade 4 to Grade 3 | 0 | 0
  HYPOGLYCEMIA Grade 4 to Grade 4 | 0 | 0

16. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Specific Thyroid Tests
Description: Blood samples were collected for conducting specific thyroid test. Baseline is defined as evaluations or events that occur before the date and time of the first dose of study treatment. Baseline was defined as evaluations or events that occur before the date and time of the first dose of study treatment or evaluations on the same date and time of the first dose of study treatment were also considered as baseline evaluations.
Time Frame: From first dose and 30 days after last dose of study therapy (Up to approximately 11 months)
Population: All treated participants with at least One on-treatment thyroid stimulating hormone (TSH) measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Docetaxel + Prednisone | Placebo + Docetaxel + Prednisone
Number analyzed (Participants) | 499 | 502
Participants
  TSH > (Upper Limit of Normal) ULN | 94 | 77
  TSH > ULN with TSH <= Upper limit of Normal (ULN) AT Baseline | 79 | 54
  TSH > ULN with at Least One FT3/FT4 Test Value < LLN | 39 | 20
  TSH > ULN With All Other FT3/FT4 Test Values >= LLN | 65 | 52
  TSH > ULN with FT3/FT4 Test Missing | 22 | 23
  TSH < Lower Limit of Normal (LLN) | 155 | 124
  TSH < LLN with TSH >= LLN at Baseline | 126 | 98
  TSH < LLN with at Least One FT3/FT4 Test Value > ULN | 33 | 14
  TSH < LLN with all other FT3/FT4 Test Values <= ULN | 116 | 106
  TSH < LLN with FT3/FT4 Test Missing | 45 | 24

17. Secondary Outcome: Time to Pain Progression as Assessed by Brief Pain Inventory-Short Form (BPI-SF)
Description: The BPI-SF is an instrument to assess pain and includes severity and interference scores. BPI-SF is an 11-item self-report questionnaire designed to assess severity and impact of pain on daily function. Participants rate severity of pain at its "worst," "least," and "average" in last 24 hours using an 11-point numerical rating scale with anchors of "no pain" and "pain as bad. The participant's assessment of pain with BPI-SF Item number 3 (pain symptoms at their worst over the last 24 hours) form basis for analysis. Time to pain progression is time between date of randomization and date of first increase in worst pain intensity. Pain progression occurred if an increase in worst pain intensity of >= 2 points is observed from baseline and maintained over 2 consecutive time periods. Baseline was evaluations or events that occur before date and time of first dose of study treatment or evaluations on same date and time of first dose of study treatment were also considered as baseline.
Time Frame: From randomization to 1st pain symptoms at their worst over the last 24 hours (Up to approximately 31 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab + Docetaxel + Prednisone | Placebo + Docetaxel + Prednisone
Number analyzed (Participants) | 514 | 516
months | 11.53 [10.28 to 13.57] | 12.42 [11.07 to 13.63]

ADVERSE EVENTS:
Time Frame: All cause mortality was collected from randomization till death (up to approximately 52 months), Serious adverse events and non-serious adverse events were collected from first dose till 100 days post last dose (Up to approximately 27 months).
Description: The number at risk for All-Cause mortality represents all randomized participants. The number at risk for serious adverse events and Other (Not Including Serious) adverse events represents all participants that received at least 1 dose of study medication.
Arm/Group | Nivolumab + Docetaxel + Prednisone | Placebo + Docetaxel + Prednisone
All-Cause Mortality (participants affected / at risk) | 259/514 | 227/516
Serious Adverse Events (participants affected / at risk) | 256/510 | 242/510
Other Adverse Events (participants affected / at risk) | 479/510 | 494/510
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Docetaxel + Prednisone (N=510) | Placebo + Docetaxel + Prednisone (N=510)
Anaemia (Blood and lymphatic system disorders) | 6 | 12
Blood disorder (Blood and lymphatic system disorders) | 0 | 1
Bone marrow infiltration (Blood and lymphatic system disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 17 | 14
Leukopenia (Blood and lymphatic system disorders) | 1 | 3
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Myelosuppression (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 9 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 2
Atrial flutter (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 3
Cardiac failure (Cardiac disorders) | 1 | 5
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Cardio-respiratory arrest (Cardiac disorders) | 3 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Immune-mediated myocarditis (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 2
Adrenal insufficiency (Endocrine disorders) | 2 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1
Immune-mediated hypophysitis (Endocrine disorders) | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 2 | 1
Cyclic vomiting syndrome (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 12 | 9
Diverticulum (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1
Enterocolitis (Gastrointestinal disorders) | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 2
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Leukoplakia oral (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 3
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3
Asthenia (General disorders) | 3 | 5
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 1
Death (General disorders) | 9 | 4
Disease progression (General disorders) | 2 | 1
Fatigue (General disorders) | 2 | 3
General physical health deterioration (General disorders) | 3 | 8
Malaise (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 2 | 2
Oedema peripheral (General disorders) | 1 | 1
Pain (General disorders) | 3 | 1
Performance status decreased (General disorders) | 1 | 0
Pyrexia (General disorders) | 7 | 3
Sudden death (General disorders) | 2 | 4
Acute cholecystitis necrotic (Hepatobiliary disorders) | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0
Biliary dilatation (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Atypical pneumonia (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 1
Bone abscess (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
COVID-19 (Infections and infestations) | 11 | 13
COVID-19 pneumonia (Infections and infestations) | 2 | 3
Cellulitis (Infections and infestations) | 4 | 2
Cellulitis streptococcal (Infections and infestations) | 1 | 0
Coronavirus infection (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 2
Device related sepsis (Infections and infestations) | 0 | 1
Diarrhoea infectious (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 3 | 1
Diverticulitis intestinal perforated (Infections and infestations) | 1 | 0
Febrile infection (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 3 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 1 | 1
Intervertebral discitis (Infections and infestations) | 1 | 0
Klebsiella urinary tract infection (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 1
Lung abscess (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 4 | 0
Oral candidiasis (Infections and infestations) | 1 | 1
Osteomyelitis (Infections and infestations) | 1 | 2
Perineal abscess (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 | 2
Pneumonia (Infections and infestations) | 18 | 8
Pneumonia aspiration (Infections and infestations) | 1 | 1
Pneumonia bacterial (Infections and infestations) | 3 | 2
Post procedural infection (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Psoas abscess (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0
Renal abscess (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Scrotal abscess (Infections and infestations) | 1 | 0
Scrotal infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 7 | 10
Septic shock (Infections and infestations) | 0 | 5
Sinusitis (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 1
Spinal cord infection (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 2
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Streptococcal infection (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 8 | 10
Urosepsis (Infections and infestations) | 2 | 2
Vascular device infection (Infections and infestations) | 1 | 2
Wound infection staphylococcal (Infections and infestations) | 0 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Chemical peritonitis (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 2 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 2
Spinal cord injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 2 | 0
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 0 | 1
General physical condition abnormal (Investigations) | 1 | 3
Hepatitis B DNA assay positive (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 2
Platelet count decreased (Investigations) | 1 | 1
Weight decreased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 4
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Immune-mediated arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Immune-mediated myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 4
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Sacral pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ependymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 | 27
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 13
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tongue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Amnesia (Nervous system disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1
Basal ganglia stroke (Nervous system disorders) | 1 | 0
Cauda equina syndrome (Nervous system disorders) | 1 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 5 | 2
Cognitive disorder (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Malignant spinal cord compression (Nervous system disorders) | 1 | 1
Nerve compression (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 6 | 6
Superior sagittal sinus thrombosis (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 1
Device dislocation (Product Issues) | 1 | 0
Device occlusion (Product Issues) | 0 | 1
Needle issue (Product Issues) | 0 | 1
Adjustment disorder with anxiety (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 4 | 5
Calculus bladder (Renal and urinary disorders) | 1 | 0
Calculus urethral (Renal and urinary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 2 | 0
Dysuria (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 13 | 2
Hydronephrosis (Renal and urinary disorders) | 0 | 2
Immune-mediated nephritis (Renal and urinary disorders) | 0 | 1
Nephritis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 2
Urethral obstruction (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 2 | 4
Urinary tract inflammation (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 2 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 13 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 8
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 1
Embolism (Vascular disorders) | 3 | 3
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Docetaxel + Prednisone (N=510) | Placebo + Docetaxel + Prednisone (N=510)
Anaemia (Blood and lymphatic system disorders) | 157 | 165
Neutropenia (Blood and lymphatic system disorders) | 40 | 58
Hypothyroidism (Endocrine disorders) | 29 | 14
Lacrimation increased (Eye disorders) | 16 | 28
Constipation (Gastrointestinal disorders) | 112 | 101
Diarrhoea (Gastrointestinal disorders) | 175 | 162
Nausea (Gastrointestinal disorders) | 108 | 134
Stomatitis (Gastrointestinal disorders) | 34 | 20
Vomiting (Gastrointestinal disorders) | 60 | 59
Asthenia (General disorders) | 113 | 108
Fatigue (General disorders) | 141 | 149
Mucosal inflammation (General disorders) | 20 | 30
Oedema peripheral (General disorders) | 90 | 108
Pain (General disorders) | 24 | 26
Pyrexia (General disorders) | 41 | 54
COVID-19 (Infections and infestations) | 63 | 62
Urinary tract infection (Infections and infestations) | 37 | 31
Infusion related reaction (Injury, poisoning and procedural complications) | 22 | 26
Alanine aminotransferase increased (Investigations) | 38 | 16
Aspartate aminotransferase increased (Investigations) | 27 | 20
Neutrophil count decreased (Investigations) | 47 | 46
Weight decreased (Investigations) | 42 | 42
White blood cell count decreased (Investigations) | 33 | 39
Decreased appetite (Metabolism and nutrition disorders) | 96 | 97
Hyperglycaemia (Metabolism and nutrition disorders) | 34 | 43
Hypocalcaemia (Metabolism and nutrition disorders) | 23 | 29
Arthralgia (Musculoskeletal and connective tissue disorders) | 84 | 97
Back pain (Musculoskeletal and connective tissue disorders) | 78 | 85
Bone pain (Musculoskeletal and connective tissue disorders) | 49 | 42
Myalgia (Musculoskeletal and connective tissue disorders) | 39 | 51
Pain in extremity (Musculoskeletal and connective tissue disorders) | 41 | 52
Dysgeusia (Nervous system disorders) | 59 | 44
Headache (Nervous system disorders) | 29 | 26
Neuropathy peripheral (Nervous system disorders) | 76 | 75
Peripheral sensory neuropathy (Nervous system disorders) | 38 | 42
Insomnia (Psychiatric disorders) | 35 | 47
Haematuria (Renal and urinary disorders) | 29 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 51 | 49
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 52 | 38
Alopecia (Skin and subcutaneous tissue disorders) | 172 | 178
Nail disorder (Skin and subcutaneous tissue disorders) | 37 | 41
Pruritus (Skin and subcutaneous tissue disorders) | 48 | 22
Rash (Skin and subcutaneous tissue disorders) | 52 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT04100018/Prot_SAP_000.pdf